CLINICAL TRIAL: NCT00670280
Title: Reducing Environmental Tobacco Smoke in NICU Infants' Homes
Brief Title: Reducing Environmental Tobacco Smoke in Neonatal Intensive Care Unit (NICU) Infants' Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Angela Stotts, Associate Professor - Family Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: R40 MC 08962-01
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Infant Environmental Tobacco Smoke Exposure
Keywords: Neonatal Intensive Care Units; Infant Morbidity; Low Birth Weight; Low Income Populations; MCH Research; Respiratory Illnesses; Substance Exposed Infants; Counseling
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention Group (Experimental): Those randomized to the Intervention group will meet twice over a two-week period with a trained counselor while visiting the neonatal intensive care unit.
  Interventions: Behavioral: Motivational Interviewing intervention
- UC Group (Active Comparator): Those randomized to the Usual Care group will receive written information on secondary smoke and infant health and will be assessed at 1 month, 3 months, and 6 months post-intervention.
  Interventions: Behavioral: Usual Care
- UC-RM Group (Active Comparator): Those randomized to the Usual Care - Reduced Measurement group will receive the same information as the Usual Care group but will be measured less often (only at 6 months post-intervention).
  Interventions: Behavioral: Usual Care - Reduced Measurement

INTERVENTIONS:
Behavioral: Motivational Interviewing intervention — Those randomized to receive the Motivational Interviewing intervention will meet twice over a two-week period with a trained counselor while visiting the neonatal intensive care unit. Each visit will consist of a 45 minute session in which household smoking practices will be assessed and discussed. Two weeks after the child has been discharged from the hospital, the counselor will contact participants via telephone for a third 20-30 minute telephone meeting. After the third contact with the counselor, a letter will be mailed to participants summarizing information covered in the three meetings.
  Arms: Intervention Group
Behavioral: Usual Care — Those randomized to receive the Usual Care intervention will receive written information on secondary smoke and infant health and will be assessed at 1 month, 3 months, and 6 months post-intervention.
  Arms: UC Group
Behavioral: Usual Care - Reduced Measurement — Those randomized to the Usual Care - Reduced Measurement intervention will receive the same written information on secondary smoke and infant health as the Usual Care intervention but will be assessed only at the 6-month timepoint.
  Arms: UC-RM Group

SUMMARY:
This study is about reducing the risks of smoke-related infant health problems. Research has shown that infants exposed to secondary smoke have higher risks of delayed lung development, respiratory illnesses, wheeze, cough, asthma, middle ear disease, and sudden infant death syndrome. Infants who have experienced low birth weight or required mechanical ventilation may be at an even greater risk for the negative effects of smoking. The purpose of this study is to evaluate the effectiveness of a 3-session program aimed at assisting the primary care giver in reducing risks to their child's health by decreasing infant smoke exposure in their home and/or reducing overall cigarette use.

Caregivers will not be required to quit smoking to take part in this program. This information will, in the future, help to identify and improve ways of reducing health problems and perhaps death in children.

DETAILED DESCRIPTION:
Approximately 38% of children aged 2 months to 5 years are exposed to environmental tobacco smoke (ETS), and compelling evidence suggests rates are even higher in low-income, less educated households. The adverse health effects of chronic ETS in children are well documented and include higher risks of delayed lung development, respiratory illnesses, wheeze, cough, asthma, middle ear disease and sudden infant death syndrome. Preterm infants admitted to a Neonatal Intensive Care Unit (NICU) are particularly vulnerable to the effects of ETS, typically exhibiting significant respiratory or chronic lung conditions prior to discharge.

The primary aim of this investigation is to develop and verify the feasibility and efficacy of a multicomponent behavioral intervention for reducing ETS exposure in a low-income, multi-ethnic population of NICU infants at particularly high social and medical risk for adverse effects of ETS. A randomized, controlled, between groups design will be used to test a hospital-based ETS reduction program based on motivational interviewing (MI). A total of 150 families with an infant at high respiratory risk in the NICU who report regular household smoking will be randomized to either MI or Usual Care. The MI intervention will include 2 one-hour counseling sessions within the 2 weeks prior to infant discharge and one telephone counseling call at two weeks post-discharge. Counseling and interviews will be conducted in Spanish or English.

The proposed research brings together highly experienced behavioral and clinical investigators, an extraordinary infrastructure, and a large population easily accessible for intervention prior to discharge. Effective brief, hospital-based interventions to reduce ETS exposure in households with NICU infants at high respiratory risk could result in substantial decreases in adverse health effects and the very large associated costs.

ELIGIBILITY:
Inclusion Criteria:

* have an infant that is 2-3 weeks prior to the estimated date of hospital discharge in the NICU at Children's Memorial Hermann Hospital
* have an infant at high respiratory risk (very low birth weight or received mechanical ventilation for >12 hours)
* report at least one person in the home who usually smokes >6 cigarettes/week in the house
* speak English or Spanish
* agree to the assessments
* attend intervention sessions (anyone who smokes in the home would be asked but not required to attend)
* live within 50 miles of our center
* have access to a telephone
* provide informed consent

Exclusion Criteria:

* severe cognitive, and/or psychiatric impairment, per judgment of NICU and research staff, that precludes cooperation with study protocol
* inability to read, write, speak English or Spanish
* inability or unwillingness to provide signed consent for participation, including parental consent if under age 18 (unless caregiver is an emancipated minor)
* inability or unwillingness to meet study requirements, including follow-up home visits for data collection purposes

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy variables will include both objective (household air nicotine levels; infant ETCO levels) and self-report measures of household ETS exposure. | 6 months post-intervention

SECONDARY OUTCOMES:
In addition to achieving lower infant smoke exposure rates in the MI condition, we expect MI will produce significant changes in several domains (e.g. self-efficacy, motivation to change). | 1 month, 3 months, and 6 months post-intervention
Additional preliminary clinical outcomes will be assessed for the generation of evidence-based hypotheses, including differential impact on respiratory symptoms and diagnoses. | 1 month, 3 months, and 6 months post-intervention
Additional preliminary clinical outcomes will be assessed for the generation of evidence-based hypotheses, including differential impact on healthcare utilization. | 1 month, 3 months, and 6 months post-intervention
Finally, the impact on ETS outcomes of having an infant with Bronchopulmonary Dysplasia will be explored. | 1 month, 3 months, and 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Stotts, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States